CLINICAL TRIAL: NCT02950025
Title: A Randomized Controlled Phase II Study of Daily Online Adaptation Versus Localization for MRI-Guided SBRT for Unresectable Primary or Oligometastatic Abdominal Malignancies
Brief Title: Daily Online Adaptation Versus Localization for MRI-Guided SBRT for Unresectable Primary or Oligometastatic Abdominal Malignancies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201611018
Record Dates: First submitted 2016-10-27; First posted 2016-10-31 (Estimated); Results first posted 2019-03-20 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-03

CONDITIONS: Pancreatic Cancer; Pancreas Cancer; Cancer of the Pancreas; Hepatocellular Carcinoma
MeSH Terms: conditions — Pancreatic Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Online non-adaptive MRI-guided SBRT (Active Comparator): * All patients will be initially planned for stereotactic body radiation therapy to a minimum dose of 50Gy in five fractions to the planning target volume (PTV)
  * Radiotherapy will consist of stereotactic body therapy, to be given over five fractions, delivered once daily or once every other day for a period of one to two weeks, for a total of five treatments
  * All patients will undergo both CT and MRI simulation in positioning appropriate for the specific treatment site
  * Quality of life questionnaire baseline, 6 weeks after treatment conclusion, and 6 months after treatment conclusion
  Interventions: Device: Online, non-adaptive MR-guided SBRT; Other: European Organization for Research and Treatment of Cancer (EORTC) QLQ-30
- Arm B: Online-Adaptive MRI-guided SBRT (Experimental): * All patients will be initially planned for stereotactic body radiation therapy to a minimum dose of 50Gy in five fractions to the planning target volume (PTV)
  * Radiotherapy will consist of stereotactic body therapy, to be given over five fractions, delivered once daily or once every other day for a period of one to two weeks, for a total of five treatments
  * All patients will undergo both CT and MRI simulation in positioning appropriate for the specific treatment site
  * When patients present for their first SBRT treatment session, the treating physician will evaluate their individual anatomy to determine if adaptive planning is indicated. Patients randomized to the online-adaptive treatment planning arm will have all tumor volumes and critical structures within 3 axial slices of the PTV re-contoured on the MR-localization image of the day
  * Quality of life questionnaire baseline, 6 weeks after treatment conclusion, and 6 months after treatment conclusion
  Interventions: Device: Online, adaptive MR-guided SBRT; Other: European Organization for Research and Treatment of Cancer (EORTC) QLQ-30

INTERVENTIONS:
Device: Online, adaptive MR-guided SBRT — Patients randomized to the online-adaptive treatment planning arm will have all tumor volumes and critical structures within 3 axial slices of the PTV re-contoured on the MR-localization image of the day. The estimated delivered dose should be calculated using the software on the console. An adapted radiation therapy plan should be generated
  Arms: Arm B: Online-Adaptive MRI-guided SBRT
Device: Online, non-adaptive MR-guided SBRT — Patients will not have online-adaptive treatment planning
  Arms: Online non-adaptive MRI-guided SBRT
Other: European Organization for Research and Treatment of Cancer (EORTC) QLQ-30 — * 30 questions
  * 28 questions about various health issues with answers ranging from 1=Not At All to 4 = Very Much
  * 1 question asking about overall health with answers ranging from 1=very poor to 7 excellent
  * 1 question asking about overall quality of life with answers ranging from 1=very poor to 7=excellent
  Other Names: EORTC QLQ-30

SUMMARY:
In light of this new technology and preliminary findings of low toxicity of online, adaptive, magnetic resonance (M)-guided stereotactic radiation on a single arm prospective study, the investigators propose to compare this technique to online MR-guided stereotactic body radiation therapy (SBRT) without adaptation. Online plan adaptation increases treatment times for patients and comprises an increased burden on technical and clinical staff. Although preliminary trial results are encouraging, it remains unclear if the dosimetric benefits of online-adaptive planning studies will translate to measurable improvements in clinical outcomes that merit its routine use. In our preliminary study, plan adaptation was most often required when tumors were adjacent to the gastrointestinal tract (the esophagus to the sigmoid colon), as those structures were most commonly the dose-limiting structures and were noted to change in location on a day-to-day basis. For these reasons, abdominal disease sites have historically highlighted the limitations of SBRT. Specifically, the investigators will enroll patients with oligometastatic or unresectable primary disease of the non-liver abdomen to a randomized, prospective trial.

Patients will be randomized to one of two treatment arms, in which they will receive either online-adaptive, MRI-guided SBRT or non-adaptive MRI-guided SBRT. Both patient groups will undergo MRI simulation and MRI treatment localization with online MR monitoring and/or gating. All patients will be treated in five fractions over one to two weeks. By adhering to strict normal tissue constraints, the investigators expect toxicity to be within the current standard of care for the non-adaptive arm, with reduction in toxicity in the arm of patients who undergo adaptation based on daily anatomic changes.

ELIGIBILITY:
Inclusion Criteria:

* Oligometastatic disease or unresectable primary abdominal malignancy with biopsy-proven primary disease histology of solid tumor categorization. Patients with a diagnosis of hepatocellular carcinoma do not require a biopsy.
* No more than three progressive sites of disease, with at least one of the disease sites to be deemed suitable for treatment with MRI-guided, online adaptive SBRT to the non-liver abdomen as per radiation oncology evaluation.
* Must be treated per protocol to lesion(s) of a single abdominal site that can reasonably be encompassed within a single treatment field. Treatment of additional site(s) outside of the abdomen while the patient is on trial is acceptable.
* The treated lesion must be within 2 cm of the abdominal gastrointestinal tract (abdominal esophagus to sigmoid colon) on the basis of cross sectional imaging study such as computed tomography (CT), positron emission tomography (PET)/CT, or MRI.
* Must be deemed medically fit for SBRT by the treating physician.
* At least 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Must have completed any systemic therapy at least one week prior to planned start of SBRT (two weeks preferred), and must have no plans to initiate systemic therapy for at least one week following end of SBRT (two weeks preferred).
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Able to understand and willing to sign an Institutional Review Board (IRB) approved, written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Primary disease of hematologic origin, lymphoma, or small cell cancer.
* Past history of external beam radiotherapy within the projected treatment field of any of the disease sites to be treated by MRI-guided, online adaptive SBRT.
* Currently receiving any other investigational agents.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Pregnant and/or breastfeeding. Patient must have a negative pregnancy test within 14 days of study entry.
* Medical contraindication to undergoing MR imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2018-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Roach, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 01/19/2017 and closed to participant enrollment on 08/13/2018.
Groups:
- Arm A: Online Non-adaptive MRI-guided SBRT: * All patients will be initially planned for stereotactic body radiation therapy to a minimum dose of 50Gy in five fractions to the planning target volume (PTV)
  * Radiotherapy will consist of stereotactic body therapy, to be given over five fractions, delivered once daily or once every other day for a period of one to two weeks, for a total of five treatments
  * All patients will undergo both CT and MRI simulation in positioning appropriate for the specific treatment site
  * Quality of life questionnaire baseline, 6 weeks after treatment conclusion, and 6 months after treatment conclusion
Period: Overall Study
Arm/Group | Arm A: Online Non-adaptive MRI-guided SBRT | Arm B: Online-Adaptive MRI-guided SBRT
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Online Non-adaptive MRI-guided SBRT | Arm B: Online-Adaptive MRI-guided SBRT | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Continuous [Median (Full Range); unit: years] | 68.5 [62 to 75] | 85 [56 to 87] | 75 [56 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 1 | 3 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Grade 3 or Greater Toxicity Occurring in Patients Receiving Online, Adaptive, MRI-guided SBRT to the Abdomen and in Patients Receiving Non-adaptive SBRT
Description: * The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.
  * Grade 3 or higher toxicities that did not predate SBRT and are probably or definitely attributable to treatment
  * Please note that the following statistical analysis was not performed due to small sample size: Statistical analysis will be powered to detect a reduction of toxicity from 35% Grade 3 or greater toxicity to 10% Grade 3 or greater toxicity using online-adaptive therapy. Statistical analysis will be one-sided test for independent proportions.
Time Frame: Up through 6 months post-treatment (approximately 6 months and 2 weeks)
Measure: Number; unit: adverse event
Arm/Group | Arm A: Online Non-adaptive MRI-guided SBRT | Arm B: Online-Adaptive MRI-guided SBRT
Number analyzed (Participants) | 2 | 3
adverse event | 0 | 1

2. Secondary Outcome: Tumor Response Rate
Description: * Tumor response rate = rate of participants who have complete or partial response at the six month follow-up
  * Complete Response (CR): Disappearance of the target lesion. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * Partial Response (PR): At least a 30% decrease in the (sum of the) diameter of the target lesion(s), taking as reference the baseline sum diameters.
Time Frame: At six month follow-up (approximately 6 months and 2 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Online Non-adaptive MRI-guided SBRT | Arm B: Online-Adaptive MRI-guided SBRT
Number analyzed (Participants) | 2 | 3
Participants | 2 | 0

3. Secondary Outcome: Progression-free Survival (PFS) Rate
Description: * PFS rate - the number of participants who have not progressed and/or died at the six-month follow-up
  * Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
  * Please note that the planned statistical analysis wasn't able to be performed due to small sample size: Utilizing Kaplan-Meier methodology
Time Frame: At six month follow-up (approximately 6 months and 2 weeks)-up
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Online Non-adaptive MRI-guided SBRT | Arm B: Online-Adaptive MRI-guided SBRT
Number analyzed (Participants) | 2 | 3
Participants | 2 | 3

4. Secondary Outcome: Disease Free Survival Rate
Description: * Disease free survival rate = the number of participants who are disease free (without any signs or symptoms of cancer) at the six-month follow-up
  * Please note that the planned statistical analysis wasn't able to be performed due to small sample size: Utilizing Kaplan-Meier methodology.
Time Frame: At six month follow-up (approximately 6 months and 2 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Online Non-adaptive MRI-guided SBRT | Arm B: Online-Adaptive MRI-guided SBRT
Number analyzed (Participants) | 2 | 3
Participants | 0 | 0

5. Secondary Outcome: Overall Survival (OS) Rate
Description: * Overall survival rate - number of participants alive at the six-month follow-up
  * Please note that the planned statistical analysis wasn't able to be performed due to small sample size: Utilizing Kaplan-Meier methodology.
Time Frame: At six month follow-up (approximately 6 months and 2 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Online Non-adaptive MRI-guided SBRT | Arm B: Online-Adaptive MRI-guided SBRT
Number analyzed (Participants) | 2 | 3
Participants | 2 | 3

6. Secondary Outcome: Patient Reported Overall Quality of Life During the Past Week as Measured by EORTC QLQ-C30 Quality of Life
Description: * Utilize both paired t-tests and repeated measures ANOVA to analyze QOL data (this was unable to be performed due to the small sample size)
  * The question asked the participant "how would you rate your quality of life during the past week?"
  * The scale ranges from 1=very poor to 7 = excellent. The higher the score the better the quality of life.
Time Frame: Pre-treatment, six-weeks post treatment, and six months post-treatment
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Arm A: Online Non-adaptive MRI-guided SBRT | Arm B: Online-Adaptive MRI-guided SBRT
Number analyzed (Participants) | 2 | 3
score on a scale
  Pre-treatment | 5 [5 to 5] | 5 [2 to 6]
  6-weeks post treatment | 6 [5 to 7] | 4 [4 to 4]
  6 months post treatment | 6 [6 to 6] | 3 [3 to 4]

7. Secondary Outcome: Number of Participants With Local Failure
Time Frame: At six month follow-up (approximately 6 months and 2 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Online Non-adaptive MRI-guided SBRT | Arm B: Online-Adaptive MRI-guided SBRT
Number analyzed (Participants) | 2 | 3
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were tracked for 6 months following the last day of SBRT. Please note, only acute adverse events were tracked. For the purposes of this protocol, adverse events collected and documented are non-hematologic acute grade 3 or higher toxicities that did not predate SBRT and are probably or definitely attributable to treatment.
Arm/Group | Arm A: Online Non-adaptive MRI-guided SBRT | Arm B: Online-Adaptive MRI-guided SBRT
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/3
Other Adverse Events (participants affected / at risk) | 0/2 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Online Non-adaptive MRI-guided SBRT (N=2) | Arm B: Online-Adaptive MRI-guided SBRT (N=3)
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Online Non-adaptive MRI-guided SBRT (N=2) | Arm B: Online-Adaptive MRI-guided SBRT (N=3)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Please note that the Principal Investigator (PI) changed for the study after all patients were off follow-up and the protocol title page didn't change at that time. This is why the listed PI is different than the PI on the title page of protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-03): https://cdn.clinicaltrials.gov/large-docs/25/NCT02950025/Prot_SAP_000.pdf